CLINICAL TRIAL: NCT04721028
Title: A Cross-sectional Study of Sarcopenia in Patients With Parkinson ' s Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021437121
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-01

CONDITIONS: Search MeSH, PubMed Database

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Body composition analysis, BMI
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Human body component analyzer — The body composition analyzer is a kind of instrument that can measure the body composition health index. It is composed of professional tester, professional consulting management software, color printer A/B machine and so on.

SUMMARY:
Parkinson's disease (PD) is the second most common neurodegenerative disease of aging. The average age of PD onset is about 60 years old. Sarcopenia is common in PD patients, and one in five Parkinson's patients is diagnosed with severe sarcopenia. The prevalence of Parkinson's disease is expected to increase in the coming decades as the population ages.

Sarcopenia is a syndrome with progressive and widespread loss of skeletal muscle mass and function, resulting in disability, loss of quality of life, and even death. Chronic disease, long-term bedridden, unreasonable diet and drug therapy may be the important factors leading to sarcopenia. China is gradually stepping into an aging society. Sarcopenia, as an age-related disease, lacks effective treatment, and has become a global public health problem and frontier research problem, bringing huge economic burden to families and society. The decline of the musculoskeletal system in the elderly will lead to muscle atrophy and loss of muscle strength, as well as decreased motor ability and balance ability, and ultimately lead to a decline in the quality of life of the elderly. The European Working Group on Sarcopenia recommends routine screening for sarcopenia in older people aged 65 and over in the community. At present, screening for sarcopenia has not received enough attention in China, and there is no unified standard for screening methods. The assessment of sarcopenia mainly focuses on three aspects: muscle mass, muscle strength and muscle function. The main symptoms of Parkinson's disease patients are postural tremor, bradykinesia and stiffness. The existence of sarcopenia may lead to poor treatment control in PD patients, and the recognition of sarcopenia in PD patients may have therapeutic effects.

This project through the cross-sectional survey of Parkinson's disease less muscle disease prevalence situation, further clear according to Parkinson's disease staging classification muscle disease prevalence, less and less by Logistic regression analysis to investigate the muscle disease and Parkinson's disease progression and the correlation between the severity of disease, for the next step nursing intervention strategies for implementation of PD patients less muscle disease provides guidance basis, to prevent and delay the less muscle disease is of great significance.

DETAILED DESCRIPTION:
The research content PD patients admitted to the Department of Neurology of our hospital from January 1, 2021 to December 31, 2022 were evaluated according to the assessment criteria for Asian sarcopenia patients (pre-sarcopenia, sarcopenia stage and severe sarcopenia stage), and the muscle mass, muscle strength and functional status of each patient were recorded. To understand the current situation of sarcopenia in PD patients, and to clarify the correlation between sarcopenia and the course and severity of disease in Parkinson's disease patients, and actively look for the influencing factors that can be intervened to guide the development of nursing intervention measures.

The research target This project through the cross-sectional survey of Parkinson's disease less muscle disease prevalence situation, further clear according to Parkinson's disease staging classification muscle disease prevalence, less and less by Logistic regression analysis to investigate the muscle disease and Parkinson's disease progression and the correlation between the severity of disease, for further implementation of PD patients with less muscle disease provide guidance on the basis of nursing intervention strategies.

The problem to be solved Dyskinesia, static tremor, and myotonia are common features of Parkinson's disease, which contribute to the loss of function and independence of Parkinson's patients. The methods used for the assessment of sarcopenia in the general population (such as the inability to measure walking speed and muscle strength) may not be applicable to PD patients, so it is necessary to consult clinical experts and teachers in the implementation process of the project.

Future research ideas

1. Through a large sample size cross-sectional survey, this project clarified the prevalence of sarcopenia in Parkinson's disease patients, collected data to clarify related preventive measures to reduce the disease burden, and provided theoretical basis for further implementation of nursing intervention strategies in the future.
2. To conduct further multicenter and cross-sectional investigation and study in the future, so as to better define the correlation between Parkinson's disease and sarcopenia.
3. To gradually develop sarcopenia assessment criteria for patients with Parkinson's disease.

1. Research method, technical route and schedule The research methods Study Design This study was a cross-sectional survey Subjects: PD patients who were admitted to the outpatient and inpatient departments of the Department of Neurology of our hospital on January 1, 2021 and December 31, 2022 were evaluated by H-Y grading scale and UPDRS-3 scale. Obtain basic patient information by consulting patient's medical records or asking patient's family members.

Included in the standard

1) Meets MDS-2015 diagnostic criteria for Parkinson's disease; 2) The patient can stand independently; 3) Informed consent of patients and their families. Exclusion criteria

1) Parkinson's disease syndrome caused by cerebrovascular diseases, encephalitis and trauma; 2) Progressive nuclear ascending paralysis, multiple system atrophy, Lewy body dementia and other Parkinson's superposition syndrome; 3) severe physical disease; 4) diseases of the digestive system; 5) wasting diseases such as infection and tumor 6) with severe mental illness or cognitive impairment. Withdrawal criteria The patient requested withdrawal. According to the literature, the incidence of sarcopenia in Parkinson's disease patients was 30.6%, the allowable error was 3%, the confidence was 0.95, and the qualified rate of the questionnaire was 90%. Combined with the above data, the sample size was calculated to be 908 cases.

Research tools and evaluation indicators Patients' basic information was obtained by consulting patients' cases or inquiring patients' family members through self-developed patients' basic information table.

1. General information: gender, age and course of disease of the patient
2. Nutrition status assessment: height, weight, triceps skin fold thickness, leg circumference, diet, MNA scale
3. Parkinson's disease symptom assessment H-Y scale, Parkinson's disease non-motor symptom rating scale (NMSS), bell drawing test
4. Patients were screened using the calf circumference and SARC-F questionnaire.<SARC-F> is a simple patient-assessed screening questionnaire, which includes 5 items in total, including strength, assisted walking, standing up, stair climbing, and the number of falls in a year. A total score of 4 or more was considered positive.

   Sarcopenia evaluation
5. Evaluation of muscle mass Bioelectrical independence analysis (BIA) was used to evaluate the patient's muscle mass (male <7.0kg/m2, female <5.7kg/m2)
6. Muscle strength assessment Hand-held gripper was used to measure the patient's main hand. When measuring grip strength, let the patient exert his hand at a constant speed to the maximum, and avoid visual feedback and verbal stimulation during exertion. Posture: 1) Standing posture: feet naturally on the ground, arms naturally droop; 2) Sitting posture: shoulder adducted neutral position, elbow flexed 90 degrees, upper arm flat with chest, forearm in neutral position; 3) Prostrate: the upper arm ababducts, the elbow is straight, and the body is 30 degrees, the forearm is neutral, the jaws up to hold the gripper, the lower end of the gripper is supported on the bed, the upper limb joints can not be flexed, moved, the gripper can not contact the body or press down.

   The AWGS 2019 recommended diagnostic threshold for grip strength for sarcopenia is less than 28.0kg for men and less than 18.0kg for women.
7. Physical function AWGS recommends the use of the 6M walking test, 5 times sitting up test to assess physical function. The time required to walk 6m at a normal pace from the beginning of the movement, without acceleration or deceleration halfway, and measured at least 2 times to record the average speed. The bound value is 1.0m/s. If the patient was unable to walk independently, a five-time sitting test was used to replace the walking test, with a threshold of ≥12s.

Data statistics

1) The prevalence of sarcopenia in PD patients was statistically analyzed; 2) The prevalence of sarcopenia in PD patients stratified by age, sex and H-Y; 3) Correlation between sarcopenia and other factors using Logistic regression model.5. Main innovations

1. Currently, there are few studies on the prevalence of sarcopenia in PD patients at home and abroad, and most of them are small sample size studies.
2. The prevalence of sarcopenia was determined according to the disease stage of PD patients.

6. Expected results and assessment indicators of the project

1. The prevalence of sarcopenia in PD patients was determined through a cross-sectional survey of outpatients with PD.
2. Logistic regression was used to analyze the correlation between sarcopenia and disease course, disease grade and other factors of Parkinson's disease, and to actively seek potential causes, especially reversible causes, so as to provide guidance for the further implementation of individualized lifestyle intervention (exercise combined nutrition) and related health education for sarcopenia.

Assessment indicators Published 1 paper in the core journal.

ELIGIBILITY:
Inclusion Criteria:

* Meets MDS-2015 diagnostic criteria for Parkinson's disease;
* The patient can stand independently;
* Informed consent of patients and their families.

Exclusion Criteria:

* Meets MDS-2015 diagnostic criteria for Parkinson's disease;
* The patient can stand independently;
* Informed consent of patients and their families.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: For PD patients who visited the outpatient and inpatient department of neurology of our hospital on January 1, 2021 and December 31, 2022,
Sampling Method: Non-Probability Sample
Enrollment: 908 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The prevalence of sarcopenia in PD patients | 2021.1-2022.12
  The prevalence of sarcopenia in PD patients was determined through a cross-sectional survey of outpatients with PD.
analyze the correlation between sarcopenia and disease course, disease grade and other factors of Parkinson's disease | 2023.1-2023.3
  Logistic regression was used to analyze the correlation between sarcopenia and disease course, disease grade and other factors of Parkinson's disease, and to actively seek potential causes, especially reversible causes, so as to provide guidance for the further implementation of individualized lifestyle intervention (exercise combined nutrition) and related health education for sarcopenia.

CONTACTS AND LOCATIONS:
Locations (1):
- SAHZhejiangU, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
The patient data will be stored in the special PD database by the researchers of this project.
  All data relating to the subject's identity will be kept confidential and will not be made public except to the extent permitted by applicable laws and/or regulations.